CLINICAL TRIAL: NCT05860972
Title: Clinical Evaluation of the Safety and Efficacy of the InMode RF Pro System With the Morpheus8 Applicator (With the 24 Pin Tip) for the Treatment of Primary Focal Hyperhidrosis of the Axillae Using Fractional RF Technology
Brief Title: Evaluation of Safety and Efficacy of Morpheus8 Applicator for the Treatment of Focal Hyperhidrosis of the Axillae Using Radio Frequency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DO611232A
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-06

CONDITIONS: Hyperhidrosis Primary Focal Axilla
Keywords: hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Intervention Model Description: Study subjects will be consecutively screened and enrolled into the study. The study will consist of an active group that will receive 2 treatments with the InMode RF Pro System with the Morpheus8 Applicator (with the 24 pin tip) and a sham group that will receive 2 sham treatments with the same InMode RF Pro System and Morpheus8 Applicator (with a sham 24 pin tip). Treatment will be performed in a preheated controlled environment (T°≥22°C). Follow up visits will occur at 1 month, 3 months, and 6 months post treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The treatments will be performed by an operator/technician who will not be blinded to the type of treatment that the subject is receiving. Objective assessment of clinical improvements such as starch-iodine tests will administered by blinded study personnel. The blinded evaluators will review photographs of the treatment areas that underwent the starch-iodine test and will be blinded as to which photos were taken at the baseline, 4-week follow-up, 12-week follow-up and 24-week follow-up visits. The HDSS, which is an objective assessment, will also be evaluated by a blinded study personnel. All subjects and study staff will be unblinded at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active group (Active Comparator): Active group that will receive 2 treatments with the InMode RF Pro System with the Morpheus8 Applicator (with the 24 pin tip)
  Interventions: Device: Morpheus8 Applicator (with the 24 pin tip) in the treatment of primary axillary hyperhidrosis.
- Sham group (Sham Comparator): Sham group that will receive 2 sham treatments with the same InMode RF Pro System and Morpheus8 Applicator (with a sham 24 pin tip).
  Interventions: Device: Morpheus8 Applicator (with the 24 pin tip) in the treatment of primary axillary hyperhidrosis.

INTERVENTIONS:
Device: Morpheus8 Applicator (with the 24 pin tip) in the treatment of primary axillary hyperhidrosis. — After subjects meet the eligibility criteria, they will be randomized with a 1:1 ratio to one of two treatment groups: Active or Sham. Subjects will receive two active or sham treatments, one month apart, with the InMode RF Pro System with the Morpheus8 Applicator and 24 pins tip and will return for three follow up visits: 4 weeks 12 weeks and 24 weeks post the second treatment

SUMMARY:
The InMode radio frequency Pro System with the Morpheus8 Applicator is a computerized system generating radio frequency energy, based on the underlying technology of Fractional RF. The Morpheus8 Applicator and 24 pin tip is used for the treatment of primary hyperhidrosis of the axillae

DETAILED DESCRIPTION:
Study subjects will be consecutively screened and enrolled into the study. The study will consist of an active group that will receive 2 treatments with the InMode radio frequency Pro System with the Morpheus8 Applicator (with the 24 pin tip) and a sham group that will receive 2 sham treatments with the same InMode radio frequency Pro System and Morpheus8 Applicator (with a sham 24 pin tip). Treatment will be performed in a preheated controlled environment (T°≥22°C). Follow up visits will occur at 1 month, 3 months, and 6 months post treatment

ELIGIBILITY:
Inclusion Criteria:

Subject is 18 years of age or older at the time of consent.

* Subject reports a quality-of-life rating of 3 or 4 on the Hyperhidrosis Disease Severity Scale (HDSS).
* Subject has primary focal axillary hyperhidrosis evidenced by at least 6 months of visible, detectable, focal, exaggerated sweating without any apparent explanation and at least two of the following:
* Bilateral and relatively symmetric
* Impairs daily activities
* Frequency of at least one episode per week
* Age of onset less than 25 years old
* Positive family history
* Cessation of focal sweating during sleep
* Subject is willing and able to comply with protocol requirements and all study visits
* Willing to have de-identified images of the treated areas taken for possible use in publications and presentations.
* Subject understands the study and has provided written informed consent

Exclusion Criteria:

Subject has secondary hyperhidrosis due to medications, infections, malignancy or endocrinopathy.

* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonal virilization.
* Severe concurrent conditions such as cardiac disorders epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Any active skin condition in the treatment area, such as sores, psoriasis, eczema and rash.
* Swollen axillary lymph nodes.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Prior endoscopic thoracic sympathectomy, liposuction or other surgery for hyperhidrosis in the treated area. Injection of botulinum toxin in the treated area within one year
* Use of Isotretinoin (Accutane®) within 6 months prior to study
* Oral anticholinergic medication use (e.g., Robinul) or cholinomimetic medication use within the last 4 weeks or planned use during the study's follow up phase.
* Currently participating in or recently participated in another clinical trial (within the last 30 days).
* History of or current neurologic deficit in the treatment limb.
* Known resistance to or history of difficulty with local anesthesia (lidocaine with epinephrine).
* Current or history of cancer, including skin cancer, or premalignant moles.
* Injury in the treatment area or any other condition that, in the opinion of the investigator, might make treatment unsafe.
* Subject has a pacemaker, defibrillator or other electronic implant anywhere in the body.
* Permanent implant in the treated area such as metal plates, screws and metal piercing or silicon.
* Females who are pregnant or nursing
* Female subjects of childbearing potential not willing to use an acceptable form of contraception for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
A statistically significant difference in the percent of responders defined as subjects reporting a Hyperhidrosis Disease Severity Scale (HDSS) score of 1 or 2 at the 4-week | 4 weeks
  A statistically significant difference in the percent of responders, defined as subjects reporting a Hyperhidrosis Disease Severity Scale (HDSS) score of 1 or 2 at the 4-week follow-up visit, in the treatment group compared to the sham group

SECONDARY OUTCOMES:
Percent of subjects with a perspiration intensity of 0-2 on the Minor's starch-iodine test Intensity | 4 weeks
  Percent of subjects with a perspiration intensity of 0-2 on the Minor's starch-iodine test Intensity Visual Scale at the 4-week follow-up visit in the treatment group compared to the sham group
Percent of responders, defined as subjects reporting a Hyperhidrosis Disease Severity Scale (HDSS) score of 1 or 2 | 12 weeks
  Percent of responders, defined as subjects reporting a Hyperhidrosis Disease Severity Scale (HDSS) score of 1 or 2 at the 12-week follow-up visit in the treatment group compared to the sham group.
Percent of subjects who achieved a 2-point or greater decline in the Hyperhidrosis Disease Severity Scale. | 4 weeks
  Percent of subjects who achieved a 2-point or greater decline in Hyperhidrosis Disease Severity Scale. from baseline at 4 weeks follow-up in the treatment group compared to the sham group

CONTACTS AND LOCATIONS:
Overall Officials: Rodney J Rohrich, MD, Principal Investigator
Locations (4):
- United States (3):
  - Skinfluence, New York, New York
  - Southeastern Dermatology, Knoxville, Tennessee
  - Dallas Plastic Surgery Institute, Dallas, Texas
- RAMBAM Medical Center, Haifa, Israel